CLINICAL TRIAL: NCT02683499
Title: A Double-blind Split-mouth Randomized Clinical Trail Evaluating Marginal Fit of Porcelain Laminate Veneers Following Finishing the Prepared Surfaces With Ultrasonic Tips Compared to the Conventional Way
Brief Title: Marginal Fit of Porcelain Veneers After Finishing Prepared Surfaces With Ultrasonic Tips
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UDDS-FixPro-01-2016
Record Dates: First submitted 2016-02-06; First posted 2016-02-17 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Tooth Discoloration
Keywords: Tooth preparation; Prosthodontics
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasonic tips (Experimental): Prepared surfaces will be finished with ultrasonic tips
  Interventions: Procedure: Ultrasonic tips
- Conventional (No Intervention): Prepared surfaces will be finished with ordinary burs

INTERVENTIONS:
Procedure: Ultrasonic tips — These tips are going to be used to give the final shape of the prepared surfaces before taking the impression for the construction of the veneers.
  Arms: Ultrasonic tips

SUMMARY:
The aim of the study is to assess the marginal fit following preparation finishing with ultrasonic tips of porcelain veneers compared to the ordinary preparation using burs only. Two-hundred and forty crowns prepared to receive porcelain veneers (in a split-mouth design). On one side of the mouth, the prepared surfaces will be finished with ultrasonic tips. Marginal fit is measured by a 'cement replica technique'.

DETAILED DESCRIPTION:
All-ceramic restoration are increasing in daily routine treatments although remain less popular than metal-ceramic crowns especially as the cost of metal rises and aesthetic requested people increases The increased demand for aesthetic treatments has led to the widespread use of metal-free ceramics for conservative restorations. Whilst studies for clinical porcelain restorations clarifies satisfactory success rates describes the reasons for failure is due to advance the techniques and materials used in dental restorations. All-ceramic restorations failures are due to several reasons, such as restoration fractures, discoloration in marginal area, marginal misfits and secondary decays. However, secondary caries is the main failure mentioned by the studies, responsible for 21% of the suddenly crown replacements. The etiology of secondary caries is as classified to primary caries, with the involvement of the same cariogenic microorganisms. The place and spread where to invade of primary and secondary lesions are also similar, with secondary caries developing mainly in the gingival tooth interface of restored teeth. Different authors have mentioned different instrumentation to prepare teeth appropriately.Preparation may be applied using diamond burs attached to sonic devices or high-speed rotating instruments with diamond or tungsten carbide burs. The action of conventional high-speed instruments applied for tooth preparation has been widely researched as well as the adhesion strengths and marginal microleakage it produces. Some authors insisted that dental surface morphology of prepared teeth is influenced by the type of bur used for preparation.

ELIGIBILITY:
Inclusion Criteria:

* aesthetic requirement with no cracks and congenital loss of any incisors.
* discolored teeth not responding to bleaching.

Exclusion Criteria:

* evidence proximal caries ,
* edge to edge occlusion
* parafunctional habits
* root canal treated teeth.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Thickness of the light silicone layer encompassed between the abutment and the veneer | measurement will be made immediately (in the same day) of applying the constructed veneers onto the prepared dental surfaces
  A light silicone material is going to be used to allow for measuring any gaps beneath the veneers. The measurement will be in micrometer using a microscope.

CONTACTS AND LOCATIONS:
Overall Officials: Anas Abdo, DDS, Principal Investigator — MSc student in Prosthodontics, University of Damascus Dental School; Mirza Allaf, DDS MSc PhD, Study Director — Associate Professor of Prosthodontics
Locations (1):
- Department of Fixed Prosthodontics, University of Damsacus, Damascus, Rif-dimashq Governorate, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayad MF. Effects of tooth preparation burs and luting cement types on the marginal fit of extracoronal restorations. J Prosthodont. 2009 Feb;18(2):145-51. doi: 10.1111/j.1532-849X.2008.00398.x. Epub 2008 Nov 18. PMID 19054303
- [Background] Ayad MF, Johnston WM, Rosenstiel SF. Influence of dental rotary instruments on the roughness and wettability of human dentin surfaces. J Prosthet Dent. 2009 Aug;102(2):81-8. doi: 10.1016/S0022-3913(09)60114-1. PMID 19643221
- [Background] Christensen RP, Ploeger BJ. A clinical comparison of zirconia, metal and alumina fixed-prosthesis frameworks veneered with layered or pressed ceramic: a three-year report. J Am Dent Assoc. 2010 Nov;141(11):1317-29. doi: 10.14219/jada.archive.2010.0076. PMID 21037189
- [Background] Eick JD, Johnson LN, Fromer JR, Good RJ, Neumann AW. Surface topography: its influence on wetting and adhesion in a dental adhesive system. J Dent Res. 1972 May-Jun;51(3):780-8. doi: 10.1177/00220345720510031401. No abstract available. PMID 4555792
- [Background] Finger WJ, Manabe A, Alker B. Dentin surface roughness vs. bond strength of dentin adhesives. Dent Mater. 1989 Sep;5(5):319-23. doi: 10.1016/0109-5641(89)90123-1. PMID 2700463
- [Background] Hickel R, Roulet JF, Bayne S, Heintze SD, Mjor IA, Peters M, Rousson V, Randall R, Schmalz G, Tyas M, Vanherle G. Recommendations for conducting controlled clinical studies of dental restorative materials. Clin Oral Investig. 2007 Mar;11(1):5-33. doi: 10.1007/s00784-006-0095-7. Epub 2007 Jan 30. PMID 17262225
- [Background] Lange RT, Pfeiffer P. Clinical evaluation of ceramic inlays compared to composite restorations. Oper Dent. 2009 May-Jun;34(3):263-72. doi: 10.2341/08-95. PMID 19544814
- [Background] Mowery AS Jr, Parker M, Davis EL. Dentin bonding: the effect of surface roughness on shear bond strength. Oper Dent. 1987 Summer;12(3):91-4. No abstract available. PMID 3306618
- [Background] Price RB, Sutow EJ. Micrographic and profilometric evaluation of the finish produced by diamond and tungsten carbide finishing burs on enamel and dentin. J Prosthet Dent. 1988 Sep;60(3):311-6. doi: 10.1016/0022-3913(88)90275-2. No abstract available. PMID 2845071